CLINICAL TRIAL: NCT00366002
Title: A 12-Week, Open-Label, Non-Randomized, Multicenter Study to Evaluate the Patient's Perception of Outcome After Treatment With Darifenacin in Overactive Bladder (OAB) Patients Dissatisfied With Prior Anticholinergic Therapy
Brief Title: Patient's Perception of Treatment Outcome With Darifenacin by Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDAR328A2404
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Overactive Bladder (OAB)
Keywords: Darifenacin,Overactive Bladder,antimuscarinic,M3 muscarinic receptor antagonist
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

ARMS (1):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin

INTERVENTIONS:
Drug: Darifenacin — Darifenacin 7,5 mg tablets once daily with the possibility to up-titrate to 15 mg once daily
  Other Names: Enablex

SUMMARY:
This study will evaluate safety, efficacy and patient's perception of outcome after treatment with darifenacin (7.5 mg once daily (o.d.) with voluntary increase up to 15 mg o.d.) in patients with OAB who are dissatisfied with prior oxybutynin extended release (ER) or tolterodine extended release (ER) therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Symptoms of OAB for at least six months prior to randomization

  * ≥ 8 micturitions on average/24 hours
  * ≥ 1 urgency episodes on average/24 hours
  * with or without UUIE

    * Patients dissatisfied with prior oxybutynin ER or tolterodine ER treatment. Patients must have been on either treatment for at least 1 week and up to 12 months preceding this study. It is required that either oxybutynin ER or tolterodine ER was the most recent OAB medication taken.
    * Patients without prior darifenacin treatment

Exclusion Criteria:

* • A mean daily urinary volume >3000 mL or a mean volume voided/micturition of >300 mL as verified in the micturition diary for two consecutive days prior to Baseline

  * Males with post-void residual (PVR) urinary volume >200 mL at Baseline
  * Clinically predominant and bothersome stress urinary incontinence, as determined by the investigator
  * Urinary retention or clinically significant bladder outlet obstruction as determined by the investigator

Other protocol-defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the patient's perception of outcome at Week 13 using the Patient Perception Bladder Condition questionnaire (PPBC).

SECONDARY OUTCOMES:
Patient's perception of outcome using the PPBC questionnaire at Week 7.
Patient's satisfaction by using the Patient Satisfaction Treatment Benefits questionnaire (PSTB, Part I) at Week 13.
Assessment of efficacy of darifenacin with respect to change from baseline in:
Number of micturitions per day at Weeks 7 and 13
Number of urgency episodes per day at Weeks 7 and 13
Number of urge urinary incontinence episodes (UUIE) per week at Weeks 7 and 13
Assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical Corporation, Study Chair — NPC
Locations (82):
- United States (82):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Chandler, Arizona
  - Investigative Site, Mesa, Arizona
  - Investigative Site, Sierra Vista, Arizona
  - Investigative Site, Tempe, Arizona
  - Investigative Site, Atherton, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Newport Beach, California
  - Investigative Site, San Diego, California
  - Investigative Site, Temecula, California
  - Investigative Site, Torrance, California
  - Investigative Site, Upland, California
  - Investigative Site, Aurora, Colorado
  - Investigative Site, Littleton, Colorado
  - Investigative Site, Wheat Ridge, Colorado
  - Investigative Site, Hollywood, Florida
  - Investigative Site, New Smyrna Beach, Florida
  - Investigative Site, Ocala, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Sarasota, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, West Palm Beach, Florida
  - Investigative Site, Weston, Florida
  - Investigative Site, Alpharetta, Georgia
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Marietta, Georgia
  - Investigative Site, Roswell, Georgia
  - Investigative Site, Snellville, Georgia
  - Investigative Site, Melrose Park, Illinois
  - Investigative Site, O'Fallon, Illinois
  - Investigative Site, Peoria, Illinois
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Greenwood, Indiana
  - Investigative Site, Topeka, Kansas
  - Investigative Site, Milford, Massachusetts
  - Investigative Site, Watertown, Massachusetts
  - Investigative Site, Flint, Michigan
  - Investigative Site, Saint Joseph, Michigan
  - Investigative Site, Chesterfield, Missouri
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Lincoln, Nebraska
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Lawrenceville, New Jersey
  - Investigative Site, West Orange, New Jersey
  - Investigative Site, Albany, New York
  - Investigative Site, Garden City, New York
  - Investigative Site, Latham, New York
  - Investigative Site, Mineola, New York
  - Investigative Site, New Hartford, New York
  - Investigative Site, Poughkeepsie, New York
  - Investigative Site, Troy, New York
  - Investigative Site, Williamsville, New York
  - Investigative Site, Burlington, North Carolina
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Concord, North Carolina
  - Investigative Site, Hickory, North Carolina
  - Investigative Site, High Point, North Carolina
  - Investigative Site, Salisbury, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Bethany, Oklahoma
  - Investigative Site, Edmond, Oklahoma
  - Investigative Site, Portland, Oregon
  - Investigative Site, Springfield, Oregon
  - Investigative Site, Pittsburgh, Pennsylvania
  - Investigative Site, Amarillo, Texas
  - Investigative Site, Corsicana, Texas
  - Investigative Site, Dallas, Texas
  - Investigative Site, Fort Worth, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Lake Jackson, Texas
  - Investigative Site, Bountiful, Utah
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Sandy City, Utah
  - Investigative Site, Richmond, Virginia
  - Investigative Site, Everett, Washington
  - Investigative Site, Lakewood, Washington
  - Investigative Site, Mountlake Terrace, Washington
  - Investigative Site, Seattle, Washington
  - Investigative Site, Vancouver, Washington
  - Investigative Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Zinner N, Kobashi K, Koochaki P, Fix D, Egermark M. Patient satisfaction with the benefits of overactive bladder treatment: exploration of influencing factors and development of a satisfaction assessment instrument. Neurourol Urodyn. 2011 Jan;30(1):62-8. doi: 10.1002/nau.20890. Epub 2010 Sep 21. PMID 20860020
- [Derived] Zinner N, Kobashi KC, Ebinger U, Viegas A, Egermark M, Quebe-Fehling E, Koochaki P. Darifenacin treatment for overactive bladder in patients who expressed dissatisfaction with prior extended-release antimuscarinic therapy. Int J Clin Pract. 2008 Nov;62(11):1664-74. doi: 10.1111/j.1742-1241.2008.01893.x. Epub 2008 Sep 22. PMID 18811599